CLINICAL TRIAL: NCT02728115
Title: First in Human Study to Evaluate Safety of Cellavita HD Investigational Product After Intravenous Application in Participants With Huntington's Disease
Brief Title: Safety Evaluation of Cellavita HD Administered Intravenously in Participants With Huntington's Disease
Acronym: SAVE-DH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: Cellavita Pesquisa Científica Ltda (Other); Azidus Brasil Scientific Research and Development Ltda (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SAVE-DH; 51005115.9.0000.5412 (Registry Identifier: CAAE)
Record Dates: First submitted 2016-03-11; First posted 2016-04-05 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Huntington Disease
Keywords: Huntington's Disease; Stem Cell; Dental Pulp Stem Cells
MeSH Terms: conditions — Huntington Disease | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cellavita HD Lower Dose (Experimental): Participants assigned to this arm will receive 3 administrations, one every 30 days, of 1x10^6 cells/weight range per administration of Cellavita HD (n= 3) .
  Interventions: Biological: Cellavita HD Lower Dose
- Cellavita HD Higher dose (Experimental): Participants assigned to this arm will receive 3 administrations, one every 30 days, of 2x10^6 cells/weight range per administration of Cellavita HD (n= 3).
  Interventions: Biological: Cellavita HD Higher dose

INTERVENTIONS:
Biological: Cellavita HD Lower Dose — The first three participants enrolled in the study will be assigned to the lower dose arm with staggered treatment, with an interval of 30 days between the first administration of the first participant and the first administration of the second participant assigned to this arm. All participants will receive a total of 3 intravenous administration, one every 30 days.
  Other Names: cellular therapy, mesenchymal stem cells
  Arms: Cellavita HD Lower Dose
Biological: Cellavita HD Higher dose — The last three participants enrolled in the study will be assigned to the higher dose arm with staggered treatment, with an interval of 30 days between the first administration of the first participant and the first administration of the second participant assigned to this arm. All participants will receive a total of 3 intravenous administration, one every 30 days.
  Other Names: cellular therapy, mesenchymal stem cells
  Arms: Cellavita HD Higher dose

SUMMARY:
Cellavita HD is a stem-cell therapy for Huntington's Disease. This is a first-in-human, non-randomized, phase I study in which participants with Huntington's Disease will receive three intravenous injections and will be followed for 5 years to evaluate safety and tolearability of product and preliminary evidence of effectiveness.

DETAILED DESCRIPTION:
This is a first-in-human, non-randomized, phase I study in which participants with HD will receive three intravenous injections of one of two doses of the investigational product, one every month for three months. Safety evaluation data will be composed by the register of adverse events (including type, frequency, intensity, seriousness, severity, and action taken related to the investigational product), could be include changes in vital signs, physical and medical evaluations, laboratory or serology tests and electrocardiogram (ECG), and by the incidence of benign and malign neoplasms. Preliminary evidence of efficacy will be evaluated by global clinical improvement (CIBIS) and evolution of disease improvement (motor, cognitive and behavioral degradation) through Unified Huntington's Disease Rating Scale - UHDRS and inflammatory markers: IL-4, IL-6, IL-10 (interleukin IL) e TNF-alpha (tumoral necrosis factor alpha). CNS improvement will be assessed by magnetic resonance imaging (MRI). Fluctuation in suicide tendency grade will be evaluated by Hamilton Depression Rating Scale (HDRS).The immunological response of HD product over the administration period will be evaluated by CD4+ and CD8+ proliferation and inflammatory markers release.

Participants who show evidence of loss of clinical benefit achieved over the course of treatment verified through worsening greater or equal to that expected for the natural course of the disease on motor, cognitive, behavioral and functional capacity symptoms assessed by the UHDRS scale, will receive additional doses of the product as long as there is clinical benefit at the Investigator's discretion and/or until the product is marketed. The same dose used by the subject during the treatment period will be administered throughout the period of additional doses.

ELIGIBILITY:
Inclusion Criteria:

* Sign and date ICF;
* Ability to follow instructions as well as ability to understand and fulfill the study requirements correctly;
* Male participant aged ≥ 21 and ≤ 65;
* Participants who submit medical report (PCR) attesting Huntington's disease with a number of CAG repeats on chromosome 4, greater than or equal to 40 and less than or equal to 50 (if the participant has not performed the examination and/or if he does not have the report available, a new exam should be done);
* Score 5 points or more in motor assessment UHDRS scale (Unified Huntington's Disease Rating Scale) at the time of enrollment;
* Score between 8 and 11 points in the functional capacity of the UHDRS scale at the time of enrollment.

Exclusion Criteria:

* Participation within 12 months in any clinical trial;
* Any medical observation data (clinical and physical) that medical research judge as a risk for subject if enrollment at the study;
* Any laboratory exam data that medical research judge as a risk for subject if enrollment at the study;
* Juvenile Huntington disease diagnosis;
* History of epilepsy;
* Diagnostic of major cognitive impairment;
* Active decompensated psychiatric disease;
* Current or prior history of neoplasia;
* Current history of gastrointestinal, hepatic, renal, endocrine, pulmonary, hematologic, immune, metabolic pathology or severe and uncontrolled cardiovascular disease;
* Diagnostic of any active infection, be it viral, bacterial, fungal, or caused by another pathogen;
* Participants who have contraindication to undergo any of the tests performed in this study, for example, have pacemakers or surgical clip;
* History of alcohol or illegal drugs abusers;
* History of 1 or more episodes of suicide in the two years before Visit V-4;
* Active smoker or have stopped smoking less than six months prior to enrollment;
* Test positive in at least one of the serological tests: HIV 1 and 2 (Anti-HIV-1,2), HTLV I and II, HBV (HBsAg, anti-HBc), HCV (anti-HCV-Ab) and VDRL (Treponema pallidum);
* History of drug allergy, including contrasts for imaging, or bovine products;
* In use or expected use of immunosuppressive drugs or prohibited medicines for the first three months after the first administration of the investigational product;
* Any clinical changes that is interpreted by the medical researcher as a risk to participant's enrollment.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Cellavita HD by periodic monitoring changes at adverse events, vital signs, laboratory tests, ECG and incidence of benign and malignant neoplasms | first year and in the following 4 years
  The safety of the investigational product will be evaluated in detail from periodic evaluations contemplating monitoring changes of:
  * Adverse events including type, frequency, intensity, seriousness, severity, and action taken related to the investigational product study;
  * Vital signs (BP, HR, axillary temperature), physical and medical examination (BMI, weight, height, medical condition - cardiovascular, pulmonary, digestive, musculoskeletal and peripheral, with emphasis on the neurological assessment and others);
  * Laboratory tests included hematologic, biochemical, urologic and serological analysis;
  * Electrocardiogram (ECG) of 12 derivations;
  * Incidence and classification of benign and malignant neoplasms in the following organs/systems: CNS, lung, liver, spleen, pancreas, prostate, testicle, urinary, hematological and skeletal system through the laboratory tests, magnetic resonance imaging, computerized tomography and ultrasonography.

SECONDARY OUTCOMES:
Preliminary efficacy of Cellavita HD by UHDRS improvement and global clinical response (CIBIS) | first year and in the following 4 years
  Will be evaluated by statistical comparison of the results of each UHDRS scale component: motor, cognitive and behavior. The global clinical response will be assessed by statistical comparison between baseline score observed by the Investigator before and after Cellavita HD treatment.
Preliminary efficacy of Cellavita HD by comparison of the inflammatory markers | first year
  Will be evaluated by statistical comparison of the inflammatory markers included IL-4, IL-6, IL-10 (interleukin IL) and TNF-alpha (tumoral necrosis factor alpha).
Immunological Response of Cellavita HD | first year
  The immunological response induced by Cellavita HD will be evaluated by statistical comparison between baseline results of CD4+ and CD8+ proliferation and the other evaluated times.
Preliminary efficacy of Cellavita HD by comparison of the CNS assessment | first year
  Will be evaluated by statistical comparison of the CNS assessment through magnetic resonance image at cortical thickness measurements, volumes of different brain structures, especially the basal ganglia, with special attention to caudate and metabolic changes identified in proton spectroscopy.
Risk of suicidal ideation by Hamilton Depression Rating Scale (HDRS) | first year and in the following 4 years
  Will be evaluated by suicidal domain. The classificatory pontuation may correspond to mild depression (score: 8 to 13), moderate depression (score: 19 - 22) and severe depression (score: > 23).

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Macedo da Silva, MD, Principal Investigator — Azidus Brasil Scientific Research and Development Ltda
Locations (1):
- Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.

REFERENCES:
- [Background] Adam OR, Jankovic J. Symptomatic treatment of Huntington disease. Neurotherapeutics. 2008 Apr;5(2):181-97. doi: 10.1016/j.nurt.2008.01.008. PMID 18394562
- [Background] Aleynik A, Gernavage KM, Mourad YSh, Sherman LS, Liu K, Gubenko YA, Rameshwar P. Stem cell delivery of therapies for brain disorders. Clin Transl Med. 2014 Jul 19;3:24. doi: 10.1186/2001-1326-3-24. eCollection 2014. PMID 25097727
- [Background] de Almeida FM, Marques SA, Ramalho Bdos S, Rodrigues RF, Cadilhe DV, Furtado D, Kerkis I, Pereira LV, Rehen SK, Martinez AM. Human dental pulp cells: a new source of cell therapy in a mouse model of compressive spinal cord injury. J Neurotrauma. 2011 Sep;28(9):1939-49. doi: 10.1089/neu.2010.1317. Epub 2011 Aug 8. PMID 21609310
- [Background] Bachoud-Levi AC, Gaura V, Brugieres P, Lefaucheur JP, Boisse MF, Maison P, Baudic S, Ribeiro MJ, Bourdet C, Remy P, Cesaro P, Hantraye P, Peschanski M. Effect of fetal neural transplants in patients with Huntington's disease 6 years after surgery: a long-term follow-up study. Lancet Neurol. 2006 Apr;5(4):303-9. doi: 10.1016/S1474-4422(06)70381-7. PMID 16545746
- [Background] Bachoud-Levi AC, Remy P, Nguyen JP, Brugieres P, Lefaucheur JP, Bourdet C, Baudic S, Gaura V, Maison P, Haddad B, Boisse MF, Grandmougin T, Jeny R, Bartolomeo P, Dalla Barba G, Degos JD, Lisovoski F, Ergis AM, Pailhous E, Cesaro P, Hantraye P, Peschanski M. Motor and cognitive improvements in patients with Huntington's disease after neural transplantation. Lancet. 2000 Dec 9;356(9246):1975-9. doi: 10.1016/s0140-6736(00)03310-9. PMID 11130527
- [Background] Ball LM, Bernardo ME, Roelofs H, van Tol MJ, Contoli B, Zwaginga JJ, Avanzini MA, Conforti A, Bertaina A, Giorgiani G, Jol-van der Zijde CM, Zecca M, Le Blanc K, Frassoni F, Egeler RM, Fibbe WE, Lankester AC, Locatelli F. Multiple infusions of mesenchymal stromal cells induce sustained remission in children with steroid-refractory, grade III-IV acute graft-versus-host disease. Br J Haematol. 2013 Nov;163(4):501-9. doi: 10.1111/bjh.12545. Epub 2013 Aug 31. PMID 23992039
- [Background] Barker RA, Mason SL, Harrower TP, Swain RA, Ho AK, Sahakian BJ, Mathur R, Elneil S, Thornton S, Hurrelbrink C, Armstrong RJ, Tyers P, Smith E, Carpenter A, Piccini P, Tai YF, Brooks DJ, Pavese N, Watts C, Pickard JD, Rosser AE, Dunnett SB; NEST-UK collaboration. The long-term safety and efficacy of bilateral transplantation of human fetal striatal tissue in patients with mild to moderate Huntington's disease. J Neurol Neurosurg Psychiatry. 2013 Jun;84(6):657-65. doi: 10.1136/jnnp-2012-302441. Epub 2013 Jan 23. PMID 23345280
- [Derived] Fernandes JMS, Pagani E, Wenceslau CV, Ynoue LH, Ferrara L, Kerkis I. A phase I, open-label study of intravenous human dental pulp stem cells (NestaCell(R)) at two dose levels in patients with Huntington's disease. Stem Cell Res Ther. 2025 Nov 4;16(1):611. doi: 10.1186/s13287-025-04703-w. PMID 41188963